CLINICAL TRIAL: NCT01145573
Title: Testing the Calcium DRI During Pregnancy: A Study of Bone Health in Black and White Women
Brief Title: Bone Health in Pregnancy
Acronym: B-Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-65
Record Dates: First submitted 2010-06-11; First posted 2010-06-16 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy
Keywords: calcium; vitamin D; bone; pregnancy
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Inactive pill taken daily
  Interventions: Dietary Supplement: Calcium or Placebo
- Calcium (Active Comparator): 1000mg of calcium taken daily
  Interventions: Dietary Supplement: Calcium or Placebo

INTERVENTIONS:
Dietary Supplement: Calcium or Placebo — Participants are randomized to take either 1000mg of calcium or placebo from week 16 of pregnancy until delivery.

SUMMARY:
Women between the ages of 18 and 45 are needed for a study that looks at the effect of calcium supplementation on bone health during pregnancy in black and white women. Study subjects will be divided into two groups. Each group will take 2 study supplements each day, the supplement will be calcium or placebo (a pill without calcium). The study involves five visits to the Children's Hospital of Oakland Research Institute; each visit will be 1-2 hours in length. There are 3 study visits during pregnancy and 2 in the first year after delivery. At each visit you will have your blood drawn and be asked questions about what you eat and what type of activities you do. At visit 16 and 36 weeks and 4 and 12 months postpartum you will have your bone density measured. You will be paid $240 for completing the study.

DETAILED DESCRIPTION:
Women between the ages of 18 and 45 are needed for a study that looks at the effect of calcium supplementation on bone health during pregnancy in black and white women. Study subjects will be divided into two groups. Each group will take 2 study supplements each day, the supplement will be calcium or placebo (a pill without calcium). The study involves five visits to the Children's Hospital of Oakland Research Institute; each visit will be 1-2 hours in length. There are 3 study visits during pregnancy and 2 in the first year after delivery. At each visit you will have your blood drawn and be asked questions about what you eat and what type of activities you do. At visit 16 and 36 weeks and 4 and 12 months postpartum you will have your bone density measured. You will be paid $240 for completing the study.

ELIGIBILITY:
Inclusion Criteria:

* First trimester of pregnancy
* Between the age of 18-45

Exclusion Criteria:

* Smoke
* Prepregnancy BMI >35
* Medical condition that will affect bone
* Takes a medication that affects bone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Peripheral cortical and trabecular bone changes during a reproductive cycle in black and white women. | 3 years

SECONDARY OUTCOMES:
Bone markers of bone formation and resorption during pregnancy and postpartum | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Fung, PhD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Childrens Hospital Oakland, Oakland, California, United States

REFERENCES:
- [Derived] Cullers A, King JC, Van Loan M, Gildengorin G, Fung EB. Effect of prenatal calcium supplementation on bone during pregnancy and 1 y postpartum. Am J Clin Nutr. 2019 Jan 1;109(1):197-206. doi: 10.1093/ajcn/nqy233. PMID 30649176